CLINICAL TRIAL: NCT04572204
Title: Management of Grades 3-5 Renal Trauma in Pediatrics: A Prospective Case Series
Brief Title: Management of Grades 3-5 Renal Trauma in Pediatrics
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdan Gameel, Resident doctor, Assiut University
Other Study IDs: Renal trauma management
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Renal Trauma
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative group
- interventional group
  Interventions: Other: Surgical

INTERVENTIONS:
Other: Surgical — Minimal: Such as PCN insertion Endosopic: Such as DJ insertion Surgical: Repair, Partial or total nephrectomy Angioembolization
  Groups: interventional group

SUMMARY:
comparing conservative management versus interventional management in hemodynamically stable paediatric patient with blunt renal trauma, evidence suggests that there is a reduced rate of renal loss and blood transfusion in patients managed conservatively.

ELIGIBILITY:
Inclusion Criteria:

* Children ( age group 0-18) who are diagnosed to have renal tissue injury grade 3-5 by contrast CT

Exclusion Criteria:

* Age group more than 18 years
* Low grade renal trauma 1-2
* Patients who get explored due to extra urologic indication without proper urologic assessment

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 60 children (age group 0-18 years) will be added to my study divided into two groups regardless of sex
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Stabilization of haemodynamic status of the patient in the first 24-72 hours | 24 to 72 hours

SECONDARY OUTCOMES:
Resolution of perinephric collection during follow up Triphasic MSCT abdomen and pelvis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided